CLINICAL TRIAL: NCT02670018
Title: A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of the Combination of Gemigliptin/Metformin HCl Sustained Release 50/2000 mg(25/1000 mg x 2 Tablets) in Comparison to Each Component Gemigliptin 50 mg and Metformin HCl Extended Release 2000 mg(1000 mg x 2 Tablets) Administered in Healthy Male Volunteers
Brief Title: BE Study of the Combinations of Gemigliptin 50mg and Metformin HCl Extended Release 2000mg in Comparison to Each Component Administered Alone
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: LG Life Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LG-DMCL005
Record Dates: First submitted 2015-12-22; First posted 2016-02-01 (Estimated); Last update posted 2016-02-02 (Estimated); Status verified 2016-01

CONDITIONS: Healthy
MeSH Terms: interventions — LC15-0444

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- G+M (Active Comparator): Coadministration of gemigliptin 50mg and metformin HCl extended release 1000mg * 2 tablets
  Interventions: Drug: gemigliptin and metformin HCl extended release
- C (Experimental): Combination of gemigliptin 25mg/metformin HCl extended release 1000mg * 2 tablets
  Interventions: Drug: gemigliptin/metformin HCl extended release

INTERVENTIONS:
Drug: gemigliptin and metformin HCl extended release — Coadministration of gemigliptin 50mg and metformin HCl extended release 1000mg * 2 tablets, for 1 day
  Arms: G+M
Drug: gemigliptin/metformin HCl extended release — Administration of combination of gemigliptin 25mg/metformin HCl extended release 1000mg * 2 tablets, for 1day
  Arms: C

SUMMARY:
A Randomized, Open-label, Single-dose, Two-way Crossover Clinical Trial to Investigate the Pharmacokinetics and Safety/Tolerability of the Combination of Gemigliptin/Metformin HCl Sustained Release 50/2000 mg(25/1000 mg x 2 tablets) in Comparison to Each Component Gemigliptin 50 mg and Metformin HCl Extended Release 2000 mg (1000 mg x 2 tablets) Administered in Healthy Male Volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Age between 19 to 45, healthy male subjects(at screening)
* Body weight between 55kg - 90kg, BMI between 18.0 - 27.0
* FPG 70-125mg/dL glucose level(at screening)
* Subject who totally understand the progress of this clinical trials, make decision by his free will, and signed a consent form to follow the progress.

Exclusion Criteria:

* Subject who has past or present history of any diseases following below.(liver including hepatitis virus carrier, kidney, Neurology,immunology,pulmonary,endocrine,hematooncology,cardiology,mental disorder.)
* Subject who had GI tract disease or(ulcer, acute or chronic pancreatitis) surgery.(appendectomy, hernioplasty are not included)
* Subject who had drug hypersensitivity reaction.(Aspirin, antibiotics)
* Subject who already participated in other trials in 3months
* Subject who had whole blood donation in 2months, or component blood donation in 1months or transfusion in 1months currently.
* Smokers.(but, if the subject did'nt smoke in 3months, can participate the trial)

Ages: 19 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2015-08; Primary Completion 2015-12 (Actual); Study Completion 2016-03 (Estimated)

PRIMARY OUTCOMES:
AUClast | up to 48h post-dose
  To evaluate AUClast of gemigliptin and metformin
Cmax | up to 48h post-dose
  To evaluate Cmax of gemigliptin and metformin

SECONDARY OUTCOMES:
Tmax of Gemigliptin, Metformin | up to 48h post-dose
AUCinf of Gemigliptin, Metformin | up to 48h post-dose
t1/2 of Gemigliptin, Metformin | up to 48h post-dose
CL/F of Gemigliptin, Metformin | up to 48h post-dose
Vd/F of Gemigliptin, Metformin | up to 48h post-dose
AUC0-48h of Gemigliptin metabolite(LC15-0636) | up to 48h post-dose
Cmax of Gemigliptin metabolite(LC15-0636) | up to 48h post-dose
Tmax of Gemigliptin metabolite(LC15-0636) | up to 48h post-dose
AUCinf of Gemigliptin metabolite(LC15-0636) | up to 48h post-dose
t1/2 of Gemigliptin metabolite(LC15-0636) | up to 48h post-dose
CL/F of Gemigliptin metabolite(LC15-0636) | up to 48h post-dose
Vd/F of Gemigliptin metabolite(LC15-0636) | up to 48h post-dose
metabolic ratio(MR) of Gemigliptin metabolite(LC15-0636) | up to 48h post-dose

CONTACTS AND LOCATIONS:
Locations (1):
- Yonsei University College of Medicine, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No